CLINICAL TRIAL: NCT02307305
Title: Does Duloxetine Reduce Chronic Pain After Total Knee Arthroplasty?
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hanyang University Seoul Hospital (Other)
Responsible Party: Principal Investigator, JIN KYU LEE, Assistant professor, Hanyang University Seoul Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: cymbaltaTKR
Record Dates: First submitted 2014-11-27; First posted 2014-12-04 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia | interventions — Duloxetine Hydrochloride; Celecoxib; Naproxen; Esomeprazole; Ultracet

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Duloxetin group (Experimental): 1. Phase I (preemptive): 2 hour before surgery (30mg for 1 day)
  2. Phase II (titration): POD#1~6 (30mg for another 6 days)
  3. Phase III (maintenance): POD#7~13(60mg for 7 days)
  4. Phase IV (tapering-1): POD#14~20 (30mg for 7 days)
  5. Phase V (tapering-2): POD#21~27 (30mg another every day for 7 days)
  plus routine pain control (celecoxib, naproxen/esomeprazole, acetaminophen/tramadol, oxycodone/naloxone)
  Interventions: Drug: Duloxetine; Drug: celecoxib, naproxen/esomeprazole, acetaminophen/tramadol, oxycodone/naloxone
- routine pain control group (Active Comparator): Preemptive analgesia : celebrex, Patient controlled analgesia (postop. 28 hours), During admission : celebrex BP or vimovo BP +ultracet ER BP, targin HS, Discharge medication: celebrex BP or vimovo BP, ultracet ER BP(PRN)
  Other name of drugs: celecoxib, naproxen/esomeprazole, acetaminophen/tramadol, oxycodone/naloxone
  Interventions: Drug: celecoxib, naproxen/esomeprazole, acetaminophen/tramadol, oxycodone/naloxone

INTERVENTIONS:
Drug: Duloxetine — 1. Phase I (preemptive): 2 hour before surgery (30mg for 1 day)
  2. Phase II (titration): POD#1~6 (30mg for another 6 days)
  3. Phase III (maintenance): POD#7~13(60mg for 7 days)
  4. Phase IV (tapering-1): POD#14~20 (30mg for 7 days)
  5. Phase V (tapering-2): POD#21~27 (30mg another every day for 7 days)
  Other Names: cymbalta
  Arms: Duloxetin group
Drug: celecoxib, naproxen/esomeprazole, acetaminophen/tramadol, oxycodone/naloxone — Preemptive analgesia : celebrex, Patient controlled analgesia (postop. 28 hours), During admission : celebrex BP or vimovo BP +ultracet ER BP, targin HS, Discharge medication: celebrex BP or vimovo BP, ultracet ER BP(PRN)
  Other Names: celebrex, vimovo, ultracet, targin

SUMMARY:
Range from 24% to 44%, with a prevalence of neuropathic-type pain from 6% to 20%-cause impairment in quality of life and functional capacity after total knee arthroplasty(TKA). Duloxetine (cymbalta) is a selective serotonin and nor-epinephrine reuptake inhibitor shown to be effective in treating chronic pain. Serotonin and norepinephrine in the brain and spinal cord are believed to both mediate core mood symptoms and help regulate the perception of pain. Its effects on depression and anxiety symptoms, as well as its effect on pain perception, may be due to increasing the activity of serotonin and norepinephrine in the central nervous system. Approved for the acute and maintenance treatment of major depressive disorder, the acute treatment of generalized anxiety disorder, the management of diabetic peripheral neuropathic pain and the management of fibromyalgia, all in adults (18+).

Investigators will compare the neuropathic pain following TKA in duloxetine group (n=84) with those in non-duloxetine group (n=84). Investigators will classify the participants in to 2 groups (duloxetine and non-duloxetine group) randomly, and primarily evaluate the degree of neuropathic pain using the S-LANSS pain scale (preoperatively and postoperatively 3 and 6 months). All participants will receive postoperative pain control after TKA using the same pain control regimen except duloxetine.

DETAILED DESCRIPTION:
Both groups of participants will receive pain control regimens as follows:

Preemptive analgesia : celebrex celecoxib, Patient controlled analgesia (postoperation 28 hours), During admission : celebrex BP or vimovo BP +ultracet ER BP, targin HS, Discharge medication: celebrex BP or vimovo BP, ultracet ER BP(PRN)

Drug generic names: celecoxib (celebrex), naproxen/esomeprazole (vimovo), acetaminophen/tramadol (ultracet ER), oxycodone/naloxone (targin)

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis of knee requiring TKA

Exclusion Criteria:

* Rheumatoid arthritis
* Other inflammatory arthritis
* Neuropsychiatric patients
* Hepatic insufficiency
* Renal insufficiency
* Patients older than 75
* Allergy or intolerance to study medications
* Patients with an ASA of IV (angina, congestive heart failure, dementia, cerebrovascular accident)
* Chronic gabapentin or pregabalin use (regular use for longer than 3 months)
* Chronic opioid use (taking opioids for longer than 3 months)

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
neuropathic pain(the self assessed-Leeds Assessment of Neuropathic Symptoms and Signs pain scale, S-LANSS) | 6 months

SECONDARY OUTCOMES:
Numeric rating scale for pain (NRS) | 6 months
American Knee Society knee and function score | 6 months
Western Ontario and McMaster University Arthritis Index (WOMAC) | 6 months
Geriatric depression scale-short form | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Choonghyeok Choi, Study Chair — Hanyang University
Locations (1):
- Department of Orthopaedic Surgery, Hanyang University, College of Medicine, Seoul, South Korea